CLINICAL TRIAL: NCT05269849
Title: Low-dose Sirolimus for Nosebleeds in HHT: a Phase II Pilot Study
Brief Title: Sirolimus for Nosebleeds in HHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Marie Faughnan, Principle Investigator, Unity Health Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200421448
Record Dates: First submitted 2022-02-14; First posted 2022-03-08 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Nosebleeds; Epistaxis
Keywords: Hereditary Hemorrhagic Telangiectasia; HHT; Sirolimus
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral sirolimus tablets (Experimental): Sirolimus starting dose of 2 mg once daily, orally adjusted as need to maintain drug blood levels of 6-10 ng/ ml The first dose will be given at the week 12 visit and participants will be observed for 30 min
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus (1, 2, or 5 mg tablets) given for 3 months followed by a washout period of 3 months

SUMMARY:
This pilot study is to determine the safety and efficacy of oral sirolimus (blood trough level 6-10ng/ml) in patients with HHT that are experiencing moderate or severe epistaxis. The effect of oral sirolimus on epistaxis will be compared to baseline using the Patient-Reported Outcome of cumulative weekly nose Bleeding Duration (PRO-CB). The PRO-CB association with biomarker variability over the duration of the study will be investigated. In the pilot study subjects will be treated with 2mg of sirolimus once daily to obtain a trough level of 6-10ng/ml for 3 months.

DETAILED DESCRIPTION:
The most common symptom of the hereditary hemorrhagic telangiectasia (HHT) disease is epistaxis. HHT is characterized by vascular (blood vessel) malformations, of the skin and mucus membranes of the nose (telangiectasia), gastrointestinal track, brain, lung and liver.

HHT is an autosomal dominant disease which is found in approximately 1 in 5000 individuals. Epistaxis affects 90% of adults with HHT, negatively affects quality of life and often causes anemia. Recent topical therapeutics trials have been negative and surgical therapies are invasive and offer only temporary benefit at best. Currently there are no highly-effective or approved systemic therapies for HHT-related epistaxis, but this is an area of active research and development. There is considerable in developing and identifying therapies that target the abnormal biology ad mechanisms in HHT, including antiangiogenic therapies, such as bevacizumab. Bevacizumab, however, is associated with significant toxicity, costly and administered intravenously.

Over the past few years, there has been considerable new evidence of the pathways involved in HHT disease and related potential therapeutic targets, including the mTOR pathway. Evidence suggests that HHT pathogenesis strongly relies on overactivated PI3K-Akt-mTOR and VEGFR2 pathways in endothelial cells. It was recently reported that the mTOR inhibitor, sirolimus, and the receptor tyrosine-kinase inhibitor, nintedanib, synergistically fully blocked, and also reversed, retinal AVMs, in the BMP9/10- immunoblocked neonatal mouse model of HHT. Subsequent unpublished preliminary data demonstrated that sirolimus was more effective than nintedanib at blocking anemia and bleeding in inducible ALK1 knockout HHT mice, and similarly effective to combined sirolimus-nintedanib. As such, sirolimus may provide therapeutic benefit for HHT patients. Human studies have shown "low-dose" sirolimus to be low risk and effective as a treatment for other vascular anomalies.

There is an urgent need for effective therapies for HHT and the chronic bleeding associated with the disease. Preliminary cellular and animal model data have identified sirolimus as a potential new pathway-based therapy in HHT. In addition, sirolimus is an interesting agent, as it is given orally and is available for repurposing. Data from other vascular malformations syndromes suggest that it can be effective in a "low-dose" range, reducing risk of toxicity, but there is only one published case report of sirolimus use in an HHT patient. This phase II pilot study will provide safety data as the primary outcome, and secondarily, efficacy data, outcome measure data and biological exploratory data, to support the planning of a future randomized and placebo -controlled clinical trial of sirolimus for epistaxis in HHT patients.

Sirolimus has been identified as a potential pathway-based therapy for HHT. Pre-clinical research has suggested that the pathogenesis of HHT is as a result of overactive mTOR and VEGFR2 pathway. Sirolimus has been found to work as an mTOR inhibitor to prevent the effects of overactive mTOR that results in arteriovenous malformations in a HHT. One clinical trial that used sirolimus to treat vascular anomalies, found that sirolimus was well tolerated and acted as an effective and safe treatment for most study participants.

Considerable experience using sirolimus in post-transplant patients and growing experience using sirolimus in patients with vascular anomalies exist. This pilot study will assess the safety and effectiveness of repurpose oral sirolimus, for epistaxis in patients with HHT.

It is hypothesized that oral sirolimus (blood trough level 6-10ng/ml) will be a safe and effective therapy for epistaxis in HHT patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Clinical HHT diagnosis (8) or genetic diagnosis of HHT
3. Epistaxis at least 15 min per week.
4. COVID-19 Vaccine (2 doses)
5. Ability to give written informed consent, including compliance with the requirements of the study.

Exclusion Criteria:

1. Allergy/intolerance to the study drug or related agents
2. Unstable medical illness
3. Acute infection
4. Creatinine > ULN (upper limit of normal)
5. Liver transaminases (AST or ALT) >= 2x ULN
6. Women participant who are pregnant or breastfeeding or plan to become pregnant during the duration of the study
7. Women of childbearing potential not on effective contraception.
8. Male participants of reproductive potential whose female partners are of childbearing potential and are not planning to use highly effective contraceptive method
9. Immunocompromised
10. History of malignancy
11. Known untreated dyslipidemia (20% above the ULN of total cholesterol and triglycerides)
12. Specific contra-indications for study drug (detailed in the product monograph)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Electrolytes | 9 months
  Sodium, potassium, chloride, total CO2
Hematology | 9 months
  Total blood count -CBC
Renal function | 9 months
  Urea, creatinine
Liver function | 9 months
  AST, ALT, total bilirubin
ferritin level | 9 months
  ferritin
Blood glucose level | 9 months
  glucose
lipid assessment | 9 months
  total cholesterol, triglycerides

SECONDARY OUTCOMES:
Epistaxis | 9 months
  Epistaxis data will be collected by PRO-CB using daily diary throughout the 9 months of the study.
Biomarkers | 9 months
  We will collect plasma for biomarkers to explore variability over time, on/off therapy and association with PRO-CB.(specific panel will be determined with the HHT Study team which may include the following: ANG2 sICAM1 PIGF TSP2 sVEGFR2, BMP9 IL6 SDF1 sVCAM1 sVEGFR3, sCD73 sIL6R TGFβ1 VEGF, sENG OPN TGFβ2 VEGF-C, GP130, PDGF-AA, sTGFβR3, VEGF-D, HGF PDGF-BB, TIMP1, sVEGFR1

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Faughnan, MD MSc FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faughnan ME, Mager JJ, Hetts SW, Palda VA, Lang-Robertson K, Buscarini E, Deslandres E, Kasthuri RS, Lausman A, Poetker D, Ratjen F, Chesnutt MS, Clancy M, Whitehead KJ, Al-Samkari H, Chakinala M, Conrad M, Cortes D, Crocione C, Darling J, de Gussem E, Derksen C, Dupuis-Girod S, Foy P, Geisthoff U, Gossage JR, Hammill A, Heimdal K, Henderson K, Iyer VN, Kjeldsen AD, Komiyama M, Korenblatt K, McDonald J, McMahon J, McWilliams J, Meek ME, Mei-Zahav M, Olitsky S, Palmer S, Pantalone R, Piccirillo JF, Plahn B, Porteous MEM, Post MC, Radovanovic I, Rochon PJ, Rodriguez-Lopez J, Sabba C, Serra M, Shovlin C, Sprecher D, White AJ, Winship I, Zarrabeitia R. Second International Guidelines for the Diagnosis and Management of Hereditary Hemorrhagic Telangiectasia. Ann Intern Med. 2020 Dec 15;173(12):989-1001. doi: 10.7326/M20-1443. Epub 2020 Sep 8. PMID 32894695
- [Background] Merlo CA, Yin LX, Hoag JB, Mitchell SE, Reh DD. The effects of epistaxis on health-related quality of life in patients with hereditary hemorrhagic telangiectasia. Int Forum Allergy Rhinol. 2014 Nov;4(11):921-5. doi: 10.1002/alr.21374. Epub 2014 Aug 21. PMID 25145809
- [Background] Whitehead KJ, Sautter NB, McWilliams JP, Chakinala MM, Merlo CA, Johnson MH, James M, Everett EM, Clancy MS, Faughnan ME, Oh SP, Olitsky SE, Pyeritz RE, Gossage JR. Effect of Topical Intranasal Therapy on Epistaxis Frequency in Patients With Hereditary Hemorrhagic Telangiectasia: A Randomized Clinical Trial. JAMA. 2016 Sep 6;316(9):943-51. doi: 10.1001/jama.2016.11724. PMID 27599329
- [Background] Shovlin CL, Guttmacher AE, Buscarini E, Faughnan ME, Hyland RH, Westermann CJ, Kjeldsen AD, Plauchu H. Diagnostic criteria for hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber syndrome). Am J Med Genet. 2000 Mar 6;91(1):66-7. doi: 10.1002/(sici)1096-8628(20000306)91:13.0.co;2-p. PMID 10751092
- [Background] Sadick H, Naim R, Sadick M, Hormann K, Riedel F. Plasma level and tissue expression of angiogenic factors in patients with hereditary hemorrhagic telangiectasia. Int J Mol Med. 2005 Apr;15(4):591-6. PMID 15754019
- [Background] Wetzel-Strong SE, Weinsheimer S, Nelson J, Pawlikowska L, Clark D, Starr MD, Liu Y, Kim H, Faughnan ME, Nixon AB, Marchuk DA. Pilot investigation of circulating angiogenic and inflammatory biomarkers associated with vascular malformations. Orphanet J Rare Dis. 2021 Sep 3;16(1):372. doi: 10.1186/s13023-021-02009-7. PMID 34479577